CLINICAL TRIAL: NCT02281851
Title: The Effects of Habitual Antioxidant Supplementation on Endogenous Antioxidants and Oxidative Damage in Well Trained Cyclists
Brief Title: Examining Endogenous Antioxidant Levels in Well Trained Cyclists
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: 125663; 13/WM/0226 (Other: NRES Committee West Midlands - Solihull)
Record Dates: First submitted 2014-10-16; First posted 2014-11-04 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Oxidative Stress
Keywords: Endogenous antioxidants; Antioxidant supplements; Vitamin Supplements; Exercise adaptations; Oxidative stress; Redox regulation; Cycling - exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Supplemented: The group consists of well-trained cyclists who habitually consume vitamin/antioxidant supplements for a period longer than 6 months
- Non-supplemented: The group consists of well-trained cyclists who do not consume vitamin/antioxidant supplements

SUMMARY:
This study will investigate whether increased habitual intake of antioxidant supplements effects the concentration of endogenous antioxidants, the response of antioxidants to exercise, and differences in oxidative damage compared to a non-supplemented group.

ELIGIBILITY:
Inclusion Criteria:

* Male,
* BMI 18.8 29.9 kg/m2
* cycle 3-7 times a week for durations longer than 60 minutes
* cycled for a minimum of 3 years
* accustomed to exhaustive cycling protocols
* healthy (no known cardiovascular or metabolic disease)

Exclusion Criteria:

* answering "NO" to any question on the general health questionnaire would result in exclusion from the study
* current participation in another clinical study
* current or recent smoker (last 30 days)
* prescription or non-prescription of anti-inflammatory use >30 days prior to the experiment commencing or any other medications that in the opinion of the investigator may interfere with redox signalling

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cyclist from the local West Midlands (United Kingdom) area will be invited to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Aldred, MSc PhD, Principal Investigator — University of Birmingham
Locations (1):
- School of Sport Exercise and Rehabilitation Sciences, University of Birmingham, Birmingham, West Midlands, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supplemented | Non-supplemented
Started | 4 | 10
Completed | 4 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supplemented | Non-Supplemented | Total
Number analyzed (Participants) | 4 | 10 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 10 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 10 | 14
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 10 | 14

OUTCOME MEASURES:

1. Primary Outcome: Difference in Resting Levels of Endogenous Antioxidant Proteins in Skeletal Muscle - Superoxide Dismutase 2 (SOD-2)
Description: To examine the effects of habitual vitamin and antioxidant supplementation on endogenous antioxidant production, participants will have a muscle biopsy taken at rest to examine any differences in endogenous antioxidant protein concentrations
Time Frame: Protein concentrations will be measured at baseline only
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Supplemented | Non-Supplemented
Number analyzed (Participants) | 4 | 10
Arbitrary Units | 0.42 (0.2) | 0.68 (0.32)

ADVERSE EVENTS:
Arm/Group | Supplemented | Non-Supplemented
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/10
Other Adverse Events (participants affected / at risk) | 0/4 | 0/10

LIMITATIONS AND CAVEATS:
We underestimated the pool of cyclists who consumed antioxidants (>6 months) and would be willing to undertake a muscle core biopsy. In addition, the vitamin supplements consumed by the participants varied in concentration, compound and variety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes